CLINICAL TRIAL: NCT01076855
Title: Guidance Programme for Elderly With Cognitive Disorders
Brief Title: Guidance for Elderly With Cognitive Disorders
Acronym: BOCS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/008
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Mild Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly with mild dementia: >70 years old and presence of a carer

SUMMARY:
The purpose of the programme is to facilitate the anticipation of dementia both in elderly patients suffering from this disease and in their carers and to diminish care burden in order to improve quality of life and daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* elderly (> 70 years) with mild dementia in presence of a carer.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly (>70 years) with mild dementia in presence of a carer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of life and care burden at 0, 3 and 6 months. | 0, 3 and 6 months

SECONDARY OUTCOMES:
Cognitive, behavioural and affective status | 0, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mirko Petrovic, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be